CLINICAL TRIAL: NCT01813149
Title: Mechanism and Treatment of Sympathetically Maintained Pain
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study halted prematurely and will not resume; participants are no longer being examined or receiving intervention. There is no data collected
Sponsor: The Cleveland Clinic (Other)
Collaborators: Murdoch University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 12-400
Record Dates: First submitted 2013-03-12; First posted 2013-03-18 (Estimated); Results first posted 2021-01-13 (Actual); Last update posted 2021-01-13 (Actual); Status verified 2020-12

CONDITIONS: Complex Regional Pain Syndrome (CRPS)
Keywords: Complex Regional Pain Syndrome (CRPS)
MeSH Terms: conditions — Complex Regional Pain Syndromes | interventions — Phenylephrine; Clonidine

STUDY DESIGN:
Intervention Model Description: This is best thought of as a single-arm study because the primary purpose for recruiting control patients is to use their skin biopsies as controls when running immunohistochemistry tests for determining α1-adrenoceptors (α1-AR) expression in CRPS patients. The primary outcomes are concerned with making comparisons between subgroups of CRPS patients, and not between CRPS patients and control patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- phenylephrine and clonidine (Experimental): Subjects will be injected with phenylephrine and clonidine at affected and unaffected sites.
  Interventions: Drug: phenylephrine and clonidine; Other: punch biopsy

INTERVENTIONS:
Drug: phenylephrine and clonidine — Subjects will be injected with phenylephrine and clonidine at both affected and unaffected sites.
Other: punch biopsy
  Other Names: After local anesthetic, subjects will receive punch biopsy (1/8"diameter and 1/8" deep) from both affected and unaffected sites.

SUMMARY:
40 CRPS patients will be recruited over a three-year period (target of 160 patients at all sites). Assessment of exclusion criteria will be undertaken during initial recruitment. Exclusion criteria are: <18 years; a second chronic pain syndrome that would interfere with pain rating; psychiatric comorbidity; pain in both hands or feet; pregnancy or breastfeeding; sympathectomy in the affected limb; use of topical medication; known sensitivity to alpha 1- adrenoceptor agonists or other contraindications. Patients will maintain their regular oral medications throughout the study period.

Assessment of sympathetically maintained pain (SMP) will require an intradermal dose of Phenylephrine to rekindle SMP and mechanical hyperalgesia. Clonidine will be used to control for affects of algometer fiction and may inhibit SMP by inhibiting the release of more norepinephrine from sympathetic nerve terminals. Skin biopsies will be obtained under sterile conditions from a site of mechanical or thermal hyperalgesia using a 3mm diameter skin biopsy punch under local anesthesia. Samples from a mirror image site on the contralateral body side will also be taken.

DETAILED DESCRIPTION:
Patients diagnosed with CRPS and control subjects will be enrolled in the study. The CRPS participants will be administered with phenylephrine (day 1) and clonidine (day 2). The control participants will not receive any intervention.

The aim of this study is to determine if expression of α1-adrenoceptors (α1-AR) altered in the skin of a subgroup of patients whose pain is associated with increased adrenergic sensitivity after nerve trauma. Increased adrenergic sensitivity will be determined by assessing pain in patients after administration of phenylephrine on day 1. Expression of α1-AR will be determined by taking skin biopsies on day 2 after administration of clonidine. Then, we will compare the expression of α1-AR in patients who were classified as having increased adrenergic sensitivity versus those who were not.

ELIGIBILITY:
Inclusion Criteria:

* CRPS patients

Exclusion Criteria:

* <18 years
* a second chronic pain syndrome that would interfere with pain rating
* psychiatric comorbidity
* pain in both hands or feet
* pregnancy or breastfeeding
* sympathectomy in the affected limb
* use of topical medication
* known sensitivity to alpha 1- adrenoceptor agonists or other contraindications

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2012-08; Primary Completion 2016-06 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- CRPS Patients: Patients diagnosed with CRPS that were enrolled in the study. The patients in this group were scheduled to be administered phenylephrine (day 1) and clonidine (day 2) in a sequential manner.
- Control Participants: Pain-free subjects (i.e. not diagnosed with CRPS) were enrolled in the study. These participants were not administered with phenylephrine or clonidine over the course of the study
Period: Overall Study
Arm/Group | CRPS Patients | Control Participants
Started | 90 | 38
Completed | 90 | 38
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- CRPS I: Patients diagnosed with CRPS I.
- CRPS II: Patients diagnosed with CRPS II. Peripheral nerve injury had been verified surgically or by a confirmatory test in 14 patients with CRPS II ("definite" nerve lesion), whereas in another 17 patients with CRPS II, a sensory examination and quantitative sensory tests indicated sensory disturbances in an anatomically plausible nerve distribution given the site and nature of the triggering event
- Control: Pain-free subjects enrolled in the study
- Total: Total of all reporting groups
Arm/Group | CRPS I | CRPS II | Control | Total
Number analyzed (Participants) | 59 | 31 | 38 | 128
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.9 (11.2) | 45.7 (10.6) | 44.4 (15.6) | 46.3 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 18 | 24 | 87
  Male | 14 | 13 | 14 | 41
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Caucasian | 58 | 31 | 38 | 127
  Race: Other | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Increased Adrenergic Sensitivity
Description: To investigate adrenergically evoked pain, 50 mg of the a1-AR agonist phenylephrine in 0.1 mL normal saline (equivalent to 2.5mMconcentration was injected intradermally into the most painful region of the dorsal and or foot and into a mirror-image site in the contralateral limb. Pain induced by the intradermal injection of phenylephrine into the contralateral limb of patients with CRPS usually resolved within 5 to 10 minutes. Therefore, pain that persisted for 15 minutes or longer (in the CRPS-affected limb) was considered to be atypical.
  Using this criterion, subjects who reported prolonged pain (a sign of adrenergic sensitivity) following the phenylephrine injection were classified as phenylephrine responders and those who didn't were classified as phenylephrine non-responders.
Time Frame: Day 1
Population: Data on pain scores were not collected from 5 CRPS patients (not administered phenylephrine [PE] per physician decision) of the initial 90 patients. Thus, data from 85 patients were analyzed. Data on control arm not reported because the only purpose for enrolling them in the trial was so that their skin biopsies could be used in immunohistochemistry analyses (see Outcome Measure 2 description). We did not plan to collect pain scores from control arm participants and they weren't administered PE.
Measure: Count of Participants; unit: Participants
Groups:
- CRPS Patients: CRPS patients who were enrolled in the study and then injected with phenylephrine
Arm/Group | CRPS Patients
Number analyzed (Participants) | 85
Participants
  Phenylephrine responders | 32
  Phenylephrine non-responders | 53

2. Primary Outcome: Expression of α1-adrenoceptors (α1-AR) in Dermal Nerve Bundles in the CRPS-affected Limb of Phenylephrine Responders and Non-responders
Description: Expression of α1-AR was determined from the skin biopsies using immunohistochemistry. Nerve bundles in the reticular dermis were identified in the affected limb of 25 patients with CRPS [only 22 of these were classified as phenylephrine responders/non-responders], in the contralateral limb of 21 patients with CRPS, and in 12 controls. Samples were processed in batches containing sections from 10 controls and from the affected and contralateral limbs of 10 patients. The α1-AR immunoreactivity (a measure of the expression of receptors) scores were transformed into standard units with a mean of 0 and a SD of 1 (ie, Z-scores). Positive scores represent greater than average α1-AR immunoreactivity (i.e. higher expression of α1-AR) compared with other samples in the run, and negative scores represent less than average α1-AR immunoreactivity. Normalized scores were averaged across multiple runs for each patient or control to obtain a mean α1-AR score.
Time Frame: Day 2, after clonidine injection
Population: After obtaining the mean α1-AR scores for all subjects at the affected/contralateral regions using the process described in the, "Outcome Measure Description", we then compared the mean α1-AR score between the subgroup of patients who were classified as either phenylephrine responders or non-responders.Skin biopsies were collected for all patients but nerve bundles in reticular dermis could only be identified in 22 phenylephrine responders/non-responders.
Measure: Mean (Standard Deviation); unit: z-score
Units Other Than Participants: CRPS-affected limbs
Groups:
- Phenylephrine Responders: CRPS-affected limbs of phenylephrine responders i.e. patients who experienced prolonged pain (>15 minutes) in the CRPS-affected limb after administration of phenylephrine
- Phenylephrine Non-responders: CRPS-affected limbs of phenylephrine non-responders i.e. patients who did not experience prolonged pain in the CRPS-affected limb after administration of phenylephrine
Arm/Group | Phenylephrine Responders | Phenylephrine Non-responders
Number analyzed (Participants) | 32 | 53
Number analyzed (CRPS-affected limbs) | 32 | 53
z-score
  Nerve bundles identified in reticular dermis: number analyzed (Participants) | 7 | 15
  Nerve bundles identified in reticular dermis: number analyzed (CRPS-affected limbs) | 7 | 15
  Nerve bundles identified in reticular dermis | 1.146 (1.009) | 0.142 (0.617)
  Nerve bundle not identified in reticular dermis: number analyzed (Participants) | 25 | 38
  Nerve bundle not identified in reticular dermis: number analyzed (CRPS-affected limbs) | 25 | 38
  Nerve bundle not identified in reticular dermis | NA (NA) — Biopsies were collected but nerve bundles in the reticular dermis could not be identified and hence α1-AR immunoreactivity could not be measured. (n=25) | NA (NA) — Biopsies were collected but nerve bundles in the reticular dermis could not be identified and hence α1-AR immunoreactivity could not be measured. (n=38)
Statistical Analysis 1: Comparison: Phenylephrine Responders vs Phenylephrine Non-responders; A t-test to see if expression of α1-AR differs between phenylephrine responders and non-responders; Test type: Superiority; p = 0.009, t-test, 2 sided; df=20 t-statistic = 2.90

3. Primary Outcome: Expression of Pain Association With Chronic Inflammation in Patients With Sympathetically Maintained Pain
Description: Determine whether heightened expression of cutaneous 1-adrenoceptors is associated with signs of chronic inflammation in patients with sympathetically maintained pain
Time Frame: Day 1
Population: Data on chronic inflammation was not collected
Groups:
- CRPS Patients: CRPS patients who were enrolled in the study and then injected with phenylephrine (on day 1) and clonidine (on day 2)
Arm/Group | CRPS Patients
Number analyzed (Participants) | 0

4. Primary Outcome: Decrease in Pain After Topical Adrenoceptor Blockade
Time Frame: 2 weeks after blockade
Population: Data were not collected--no patients were given a topical adrenoreceptor antagonist.
Groups:
- CRPS Patients: CRPS patients who were enrolled in the study and then administered with a topical adrenoreceptor antagonist
Arm/Group | CRPS Patients
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: Adverse events are reported for each intervention. Of the 90 CRPS patients scheduled to received phenylephrine and clonidine, 5 weren't administered any due to physician decision.
Groups:
- Phenylephrine: CRPS Patients: CRPS patients who were enrolled in the study and then administered phenylephrine (Day 1)
- Clonidine: CRPS Patients: CRPS patients who were enrolled in the study and then administered clonidine (Day 2)
- CRPS Patients: CRPS patients who were enrolled in the study but did not receive phenylephrine or clonidine.
- Control: Participants who were not diagnosed with CRPS and were not administered either phenylephrine or clonidine
Arm/Group | Phenylephrine: CRPS Patients | Clonidine: CRPS Patients | CRPS Patients | Control
All-Cause Mortality (participants affected / at risk) | 0/85 | 0/85 | 0/5 | 0/38
Serious Adverse Events (participants affected / at risk) | 0/85 | 0/85 | 0/5 | 0/38
Other Adverse Events (participants affected / at risk) | 0/85 | 0/85 | 0/5 | 0/38

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No